CLINICAL TRIAL: NCT02986880
Title: A Dose-response, Randomized, Double-blind Study to Evaluate the Effect of Type-A Botulinum Toxin in the Post-radiosurgical Neck Contractures
Brief Title: Effect of Type-A Botulinum Toxin in the Post-radiosurgical Neck Contractures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011/08; 2011-000889-35 (EudraCT Number)
Record Dates: First submitted 2016-12-06; First posted 2016-12-08 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Cervical Spasm; Radiotherapy Side Effect; Botulinum Toxin
MeSH Terms: conditions — Radiation Injuries | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (10):
- Group D1 (Experimental): Patients receiving the toxin in SCM and the placebo in trapezius muscle and splenius capitis. Patients receiving the dose of 30 units (U) at injection point, totalling 120 U.
  Interventions: Drug: Botulinum toxin A
- Group D2 (Experimental): Patients receiving the toxin in the SCM and the placebo in the trapezius muscle and the splenius capitis. Patients receiving the dose of 60 units (U) at injection point, totalling 240 U.
  Interventions: Drug: Botulinum toxin A
- Group D3 (Experimental): Patients receiving the toxin in the SCM and the placebo in the trapezius muscle and the splenius capitis. Patients receiving the dose of 100 units (U) at injection point, totalling 400 U.
  Interventions: Drug: Botulinum toxin A
- Group A1 (Experimental): Patients receiving the toxin in trapezius muscle and splenius capitis and the placebo in SCM . Patients receiving the dose of 30 units (U) at injection point, totalling 180 U.
  Interventions: Drug: Botulinum toxin A
- Group A2 (Experimental): Patients receiving the toxin in trapezius muscle and splenius capitis and the placebo in SCM . Patients receiving the dose of 60 units (U) at injection point, totalling 360 U.
  Interventions: Drug: Botulinum toxin A
- Group A3 (Experimental): Patients receiving the toxin in trapezius muscle and splenius capitis and the placebo in SCM . Patients receiving the dose of 100 units (U) at injection point, totalling 600 U.
  Interventions: Drug: Botulinum toxin A
- Group F1 (Experimental): Patients receiving the toxin in the third muscles groups. Patients receiving the dose of 30 units (U) at injection point, totalling 300 U.
  Interventions: Drug: Botulinum toxin A
- Group F2 (Experimental): Patients receiving the toxin in the third muscles groups. Patients receiving the dose of 60 units (U) at injection point, totalling 600 U.
  Interventions: Drug: Botulinum toxin A
- Group F3 (Experimental): Patients receiving the toxin in the third muscles groups. Patients receiving the dose of 100 units (U) at injection point, totalling 1000 U.
  Interventions: Drug: Botulinum toxin A
- Group P (Placebo Comparator): Patients receiving placebo in the third muscles groups
  Interventions: Procedure: Placebo

INTERVENTIONS:
Drug: Botulinum toxin A
  Arms: Group A1; Group A2; Group A3; Group D1; Group D2; Group D3; Group F1; Group F2; Group F3
Procedure: Placebo — Injection of sodium chloride (NaCl) 9/1000
  Arms: Group P

SUMMARY:
The main objective of the study is to estimate the efficiency and to determine the optimal dose of Botulinum toxin A, administered by intramuscular way in cervical spasms after radiotherapy, as well as the optimal sites for these injections.

The concerned muscular groups are the sternocleidomastoid (SCM), the trapezius muscle and the splenius capitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 18 to 75 years old;
* malignant Tumor of aerodigestive ways, in forgiveness;
* Treatment containing the external radiotherapy ended since > 6 months
* Life expectancy > 6 months;
* patient complaining from cervical spasms with functional disability;
* Negative Pregnancy test;
* Women under effective contraception;
* Patients benefiting from a national insurance scheme;
* Patient having given a written consent.

Exclusion Criteria:

* Cervico-facial Surgery with reconstruction by pedicled flap
* Implantable Chamber with catheter in the internal jugular vein near the spasm;
* Muscular, neurological Pathology or malformative pulling a disorder of perception of the pain, an amyotrophy, a muscular weakness affecting the cervical axis or the upper limbs;
* Disorder generalized by the muscular activity (ex myasthenia);
* Cervical osseous or muscular Pathology pulling pains and disability before the beginning of the treatment (cervical degenerative osteoarthritis diagnosed to the cervical radiography, the slipped disc);
* Previous cervical injection of botulinum toxin ;
* Local Infection at the level of one of the sites proposed for injection;
* Histories of epilepsy;
* Patients presenting a hypersensitivity to the botulinum neurotoxin A or in one of its excipients;
* Patients under anticoagulation therapy, Under antibiotic treatment by aminoglycosides or amino 4 quinoline, under myorelaxant treatment or that must undergo an intervention with curarisation;
* Patients for whom a surgical operation is planned in the zone interested in the treatment
* Pregnant or breast-feeding Women;
* Patients for whom questionnaires will not be assessable (handicaps of communication, patient not speaking French, etc.).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-06; Primary Completion 2014-01-10 (Actual); Study Completion 2014-01-10 (Actual)

PRIMARY OUTCOMES:
Cervical mobility degree | 6 months

SECONDARY OUTCOMES:
Quality of Life Questionnaire Module for Head and Neck Cancer (QLQ-H&N35) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Christine Bach, Principal Investigator — Hopital Foch
Locations (1):
- Hopital Foch, Suresnes, France

IPD SHARING:
Plan to Share IPD: No